CLINICAL TRIAL: NCT07249489
Title: A First in Human (FIH) Early Feasibility Study (EFS) to Evaluate the Safety and Performance of the Nanochon Chondrograft™ Implant for Re-surfacing of Cartilage Lesions
Brief Title: Nanochon Chondrograft First in Human (FIH) Early Feasibility Study (EFS) - Canada
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanochon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-2024-CAN
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Knee Cartilage Lesions
Keywords: Knee cartilage lesions; Medial femoral condyle lesion; Lateral femoral condyle lesion; Trochlea articular cartilage lesion

STUDY DESIGN:
Intervention Model Description: All participants will undergo a mini arthrotomy or arthroscopic surgical implantation of the Nanochon Chondrograft
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nanochon Chondrograft (Experimental): Mini arthrotomy or arthroscopic surgical implantation of the Nanochon Chondrograft
  Interventions: Device: Nanochon Chondrograft

INTERVENTIONS:
Device: Nanochon Chondrograft — Mini arthrotomy or arthroscopic surgical implantation of the Nanochon Chondrograft

SUMMARY:
The goal of this First in Human study is to learn if the Nanochon Chondrograft Implant is a safe primary surgical treatment for participants with cartilage lesions in the knee. This study will include males and females between the ages of 22 and 60.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥22 years and ≤ 60 years of age
* MRI knee evaluation completed within 6 months prior to enrollment
* Participant must be able to read and speak English
* Participant must voluntarily sign the REB approved informed consent form (ICF)

Exclusion Criteria:

* Any known systemic cartilage and/or bone disorder, such as, but not limited to, osteoporosis, chondrodysplasia or osteogenesis imperfecta
* Requires bilateral knee surgery
* Pregnancy, planning to become pregnant or breast feeding
* Any significant illness (metastasis cancer of any type) that decreases the probability of the participant's survival to 12 months
* Known insulin dependent diabetes mellitus
* Steroid treatment (oral or IV) within the past 6 months
* Participant is:

  1. receiving workman's compensation
  2. receiving prescription narcotic medication
  3. active with litigation relating to musculoskeletal injuries or disorders
  4. a prisoner or pending incarceration
* Comorbidities that could impact study participation or results (e.g., autoimmune disorder, HIV, neuropathic pain or fibromyalgia, restless leg syndrome, active infection, or pain requiring chronic pain management), in the opinion of the investigator at the time of enrollment
* Significant psychiatric disorders (e.g., major depression, anxiety disorders, bipolar disorder, and schizophrenia)
* Substance and/or alcohol dependence and/or abuse based on clinical history, physical exam and participant presentation
* Current participation in another drug or device study that, in the opinion of the investigator at the time of enrollment, would interfere with participation in this study
* Participant has claustrophobia or implanted metallic devices (e.g., cardiac pacemakers, insulin pumps, nerve stimulators), medically implanted clips or other electronically, magnetically or mechanically activated implants that would contraindicate undergoing an MRI
* Known allergy or hypersensitivity to any investigational device materials.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Device Event Effects | Month 12
  Absence of Serious Adverse Device Event Effects (SADEs) through Month 12

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Fraser Orthopaedic Institute, New Westminster, British Columbia
  - University of British Columbia, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time.